CLINICAL TRIAL: NCT05596734
Title: A PHASE 1/2 STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF COMBINED MODIFIED RNA VACCINE CANDIDATES AGAINST COVID-19 AND INFLUENZA IN HEALTHY INDIVIDUALS
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of Combined Modified RNA Vaccine Candidates Against COVID-19 and Influenza
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C5261001; NCT05596734 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-10-26; First posted 2022-10-27 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Influenza, Human; COVID-19
Keywords: SARS-Cov-2; COVID-19; Influenza; Grippe; Flu; Vaccine; RNA vaccine
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Masking Description: Substudy A: Open-label unblinded.
  Substudy B: Participants are blinded to their assigned study intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (18):
- SSA: qIRV + bivalent BNT162b2 (dose level combination 1) (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSA: qIRV + bivalent BNT162b2 (dose level combination 2) (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSA: qIRV + bivalent BNT162b2 (dose level combination 3) (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSA: qIRV (dose level 1) (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: qIRV (22/23)
- SSA: qIRV (dose level 2) (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: qIRV (22/23)
- SSA: bivalent BNT162b2 (dose level 1) + QIV (Experimental): BNT162b2 administered intramuscularly into the deltoid muscle of the right arm, QIV administered intramuscularly into the deltoid muscle of the left arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: QIV
- SSB: QIV + bivalent BNT162b2 (original/Omi BA.4/BA.5) (Experimental): BNT162b2 administered intramuscularly into the deltoid muscle of the right arm, QIV administered intramuscularly into the deltoid muscle of the left arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: QIV
- SSB: QIV + bIRV/bivalent BNT162b2 (original/Omi BA.4/BA.5) (Experimental): BNT162b2 administered intramuscularly into the deltoid muscle of the right arm, QIV administered intramuscularly into the deltoid muscle of the left arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: QIV; Biological: bIRV
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 1 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 2 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 3 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 4 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 5 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 6 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 7 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 8 (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: qIRV (22/23)
- SSB: tIRV/bivalent BNT162b2(original/Omi\BA.4/BA.5) (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5); Biological: tIRV
- SSB: qIRV (Experimental): Administered intramuscularly into the deltoid muscle of the right arm
  Interventions: Biological: qIRV (22/23)

INTERVENTIONS:
Biological: bivalent BNT162b2 (original/Omi BA.4/BA.5) — Intramuscular injection
  Arms: SSA: bivalent BNT162b2 (dose level 1) + QIV; SSA: qIRV + bivalent BNT162b2 (dose level combination 1); SSA: qIRV + bivalent BNT162b2 (dose level combination 2); SSA: qIRV + bivalent BNT162b2 (dose level combination 3); SSB: QIV + bIRV/bivalent BNT162b2 (original/Omi BA.4/BA.5); SSB: QIV + bivalent BNT162b2 (original/Omi BA.4/BA.5); SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 1; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 2; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 3; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 4; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 5; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 6; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 7; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 8; SSB: tIRV/bivalent BNT162b2(original/Omi\BA.4/BA.5)
Biological: qIRV (22/23) — Intramuscular injection
  Arms: SSA: qIRV (dose level 1); SSA: qIRV (dose level 2); SSA: qIRV + bivalent BNT162b2 (dose level combination 1); SSA: qIRV + bivalent BNT162b2 (dose level combination 2); SSA: qIRV + bivalent BNT162b2 (dose level combination 3); SSB: qIRV; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 1; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 2; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 3; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 4; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 5; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 6; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 7; SSB: qIRV/bivalent BNT162b2 (original/ Omi BA.4/BA.5) at dose-level combination 8
Biological: QIV — Intramuscular injection
  Arms: SSA: bivalent BNT162b2 (dose level 1) + QIV; SSB: QIV + bIRV/bivalent BNT162b2 (original/Omi BA.4/BA.5); SSB: QIV + bivalent BNT162b2 (original/Omi BA.4/BA.5)
Biological: bIRV — Intramuscular injection
  Arms: SSB: QIV + bIRV/bivalent BNT162b2 (original/Omi BA.4/BA.5)
Biological: tIRV — Intramuscular injection
  Arms: SSB: tIRV/bivalent BNT162b2(original/Omi\BA.4/BA.5)

SUMMARY:
Substudy A: This is a Phase 1 randomized, open-label study to describe the safety and immunogenicity of up to 3 dose- level combinations of modRNA quadrivalent influenza vaccine (qIRV (22/23)) and bivalent BNT162b2 (original/Omi BA.4/BA.5). Participants will receive either:

* qIRV (22/23)/bivalent BNT162b2 (original/Omi BA.4/BA.5), at 1 of the 3 dose-level combinations
* qIRV (22/23) at dose level 1,
* qIRV (22/23) at dose level 2, or
* bivalent BNT162b2 (original/Omi BA.4/BA.5) at dose level 1 administered concurrently in the opposite arm to commercially licensed quadrivalent influenza vaccine (QIV).

Substudy B: This Phase 1/2 study will describe the safety, tolerability, and immunogenicity of quadrivalent influenza vaccine (qIRV)/bivalent BNT162b2 (original/Omi BA.4/BA.5), trivalent influenza vaccine (tIRV)/bivalent BNT162b2 (original/Omi BA.4/BA.5), and bivalent influenza vaccine (bIRV)/bivalent BNT162b2 (original/Omi BA.4/BA.5) when given concurrently with licensed quadrivalent influenza vaccine (QIV).

ELIGIBILITY:
SSA: Inclusion Criteria:

* Male or female participants 18 years of age and older
* Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent as described in the protocol.
* For participants 18 through 64 years of age: participants who have received 3 prior doses of 30 µg BNT162b2, with the last dose being 150 to 365 days before Visit 1 (Day 1).
* For participants 65 years of age and older: participants who have received 4 or 5 prior doses of a modRNA SARS-CoV-2 vaccine, with the last dose being a bivalent vaccine, 120 days to 365 days before Visit 1 (Day 1).
* For Participants 65 years of age and older: receipt of licensed influenza vaccination for the 2022-2023 northern hemisphere season 120 days or more before study intervention administration.

SSA: Exclusion Criteria:

* History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency.
* Bleeding diathesis or condition associated with prolonged bleeding.
* Women who are pregnant or breastfeeding.
* Allergy to egg proteins (egg or egg products) or chicken proteins.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before enrollment through conclusion of the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or planned receipt throughout the study.
* For participants 18 through 64 years of age: vaccination with any investigational or licensed influenza vaccine within 6 months (175 days) before study intervention administration.
* Participation in other studies involving a study intervention within 28 days before randomization. Anticipated participation in other studies within 28 days after receipt of study intervention in this study.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
* Participation in strenuous or endurance exercise through Visit 3 of the study.
* Prior history of heart disease.
* Any abnormal screening troponin I laboratory value.
* Screening 12-lead ECG that, as judged by the investigator, is consistent with probable or possible myocarditis or pericarditis, or demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.

SSB: Inclusion Criteria

* Male or female participants 18 years of age and older
* Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
* Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
* Capable of giving signed informed consent as described in the protocol.
* Participants who have received at least 3 prior US-authorized mRNA COVID-19 vaccines, with the last dose being an updated (bivalent) vaccine given at least 150 days before Day 1.

SSB: Exclusion Criteria

* Medical or psychiatric condition, including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality, that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
* Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
* Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate intramuscular injection
* Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before enrollment through conclusion of the study.
* Receipt of blood/plasma products, immunoglobulin, or monoclonal antibodies, from 60 days before study intervention administration, or planned receipt throughout the study.
* Vaccination with any investigational or licensed influenza vaccine within 6 months (175 days) before study intervention administration, or ongoing receipt of chronic antiviral therapy with activity against influenza
* Participation in other studies involving administration of a study intervention within 28 days prior to, and/or during, participation in this study.
* Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.
* Initial enrollment only: Participation in strenuous or endurance exercise through Visit 3 (initial enrollment phase).
* Initial enrollment only: Prior history of heart disease of concern
* Initial enrollment only: Screening 12-lead ECG that, as judged by the investigator, is consistent with probable or possible myocarditis or pericarditis, or demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1019 (Actual)
Dates: Start 2022-10-28 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2023-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (57):
- United States (57):
  - North Alabama Research Center, Athens, Alabama
  - The Heart Center, Athens, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - The Pain Center of Arizona, Phoenix, Arizona
  - Orange County Research Center, Lake Forest, California
  - Orange County Heart Institute, Orange, California
  - California Research Foundation, San Diego, California
  - Orange County Research Center, Tustin, California
  - Proactive Clinical Research,LLC, Fort Lauderdale, Florida
  - Finlay Medical Research, Greenacres City, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Research Centers of America ( Hollywood ), Hollywood, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Gerardo Polanco, MD, Miami, Florida
  - Research Institute of South Florida, Miami, Florida
  - Entrust Clinical Research, Miami, Florida
  - Jackson Medical Group Cardiac Care, Miami, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - United Medical Research, Port Orange, Florida
  - Velocity Clinical Research, Savannah, Savannah, Georgia
  - Savannah Medical Group, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Great Lakes Clinical Trials - Ravenswood, Chicago, Illinois
  - Retina Associates, Elmhurst, Illinois
  - Affinity Health, Oak Brook, Illinois
  - Alliance for Multispecialty Research, LLC, Oak Brook, Illinois
  - Alliance for Multispecialty Research, LLC, Wichita, Kansas
  - Jadestone Clinical Research, Silver Spring, Maryland
  - Michigan Center of Medical Research (MICHMER), Farmington Hills, Michigan
  - Pradeep Chandra, DO, FACC, Bridgeton, Missouri
  - Clinical Research Professionals, Chesterfield, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Pioneer Heart Institute, Lincoln, Nebraska
  - Quality Clinical Research, Omaha, Nebraska
  - Velocity Clinical Research, Omaha, Omaha, Nebraska
  - ActivMed Practices & Research, LLC., Portsmouth, New Hampshire
  - SUNY Upstate Medical University Institute for Global Health, Syracuse, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Main Street Physician's Care, Little River, South Carolina
  - McLeod Cardiology Associates - Little River, Little River, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - DM Clinical Research, Martin Diagnostic Clinic, Tomball, Texas
  - DM Clinical Research, Tomball, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5261001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 2 sub studies: Sub study A and Sub study B. A total of 1019 participants were enrolled, out of which 1009 participants were vaccinated (sub study A: 377 and sub study B: 632).
Pre-assignment Details: Interventions administered: quadrivalent influenza modRNA vaccine (qIRV), trivalent influenza modRNA vaccine (tIRV), Bivalent BNT162b2 (Original/Omi BA.4/BA.5) and quadrivalent influenza vaccine (QIV).
Groups:
- Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 1- 90 mcg) (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg: Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 60 mcg (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 2- 90 mcg) (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy A, 18-64 Years: qIRV 30 mcg; Substudy B, 18-64 Years: qIRV (30 mcg): Participants aged 18-64 years were administered qIRV 30 mcg intramuscularly on Day 1.
- Substudy A, 18-64 Years: qIRV 60 mcg: Participants aged 18-64 years were administered qIRV 60 mcg intramuscularly on Day 1.
- Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV: Participants aged 18-64 years were administered Bivalent BNT162b2 30 mcg (Original/OMI BA.4/BA.5) and concurrent administration of licensed QIV in opposite arm intramuscularly on Day 1. Dose strength for licensed QIV was not disclosed as it acted as comparator and was administered per local regulations.
- Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1): Participants aged greater than or equal to (>=) 65 years were administered qIRV and Bivalent BNT162b2 (Combination 1- 90 mcg) (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg: Participants aged >=65 years were administered qIRV and Bivalent BNT162b2 60 mcg (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2): Participants aged >=65 years were administered qIRV and Bivalent BNT162b2 (Combination 2- 90 mcg) (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy A, >=65 Years: qIRV 30 mcg: Participants aged >=65 years were administered qIRV 30 mcg intramuscularly on Day 1.
- Substudy A, >=65 Years: qIRV 60 mcg: Participants aged >=65 years were administered qIRV 60 mcg intramuscularly on Day 1.
- Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV: Participants aged >=65 years were administered Bivalent BNT162b2 30 mcg (Original/OMI BA.4/BA.5) and concurrent administration of licensed QIV in opposite arm intramuscularly on Day 1. Dose strength for licensed QIV was not disclosed as it acted as comparator and was administered per local regulations.
- Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg): Participants aged 18-64 years were administered bivalent BNT162b2 30 mcg (Original/OMI BA.4/BA.5) and licensed QIV concurrently in opposite arm intramuscularly on Day 1. Dose strength for licensed QIV was not disclosed as it acted as comparator and was administered per local regulations.
- Substudy B, 18-64 Years: QIV and bIRV/Bivalent BNT162b2 (45 mcg): Participants aged 18-64 years were administered bIRV and Bivalent BNT162b2 45 mcg (OMI BA.4/BA.5) and licensed QIV concurrently in opposite arm intramuscularly on Day 1. Dose strength for licensed QIV was not disclosed as it acted as comparator and was administered per local regulations.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 1- 90 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 2- 90 mcg)(OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (60 mcg Combination 1): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 1- 60 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 75 mcg (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (90 mcg Combination 3): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 3- 90 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (60 mcg Combination 2): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 2- 60 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 4- 90 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 3- 60 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg): Participants aged 18-64 years were administered tIRV and Bivalent BNT162b2 75 mcg (OMI BA.4/BA.5) intramuscularly on Day 1.
Period: Substudy A
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV/Bivalent BNT162b2 (45 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Started ((as vaccinated)) | 30 | 28 | 30 | 30 | 30 | 32 | 33 | 32 | 33 | 33 | 33 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 28 | 28 | 29 | 30 | 30 | 32 | 32 | 32 | 33 | 33 | 33 | 33 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Substudy B
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV/Bivalent BNT162b2 (45 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV/Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Started ((as vaccinated)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 29 | 32 | 124 | 122 | 114 | 31 | 30 | 33 | 30 | 26 | 32 | 29
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 27 | 32 | 122 | 118 | 112 | 30 | 28 | 33 | 30 | 26 | 32 | 28
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 4 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received the study intervention. Participants were analyzed according to the treatment which they received.
Groups:
- Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg): Participants aged >=65 years were administered qIRV and Bivalent BNT162b2 60 mcg (original/OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg): Participants aged 18-64 years were administered bIRV and Bivalent BNT162b2 45 mcg (OMI BA.4/BA.5) and licensed QIV concurrently in opposite arm intramuscularly on Day 1. Dose strength for licensed QIV was not disclosed as it acted as comparator and was administered per local regulations.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 2- 90 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 1- 60 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 3- 90 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2): Participants aged 18-64 years were administered qIRV and Bivalent BNT162b2 (Combination 2- 60 mcg) (OMI BA.4/BA.5) intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg) | Total
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32 | 33 | 32 | 33 | 33 | 33 | 33 | 29 | 32 | 124 | 122 | 114 | 31 | 30 | 33 | 30 | 26 | 32 | 29 | 1009
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (11.68) | 44.4 (12.75) | 43.1 (12.45) | 42.9 (10.53) | 46.2 (11.78) | 40.5 (12.70) | 71.5 (5.33) | 71.2 (5.53) | 71.4 (4.32) | 70.8 (4.27) | 71.6 (4.55) | 71.7 (4.67) | 40.9 (11.99) | 44.1 (12.86) | 46.4 (12.13) | 45.9 (12.56) | 44.9 (14.25) | 47.0 (11.64) | 48.6 (10.17) | 47.1 (11.79) | 47.9 (9.75) | 46.9 (12.96) | 46.0 (11.93) | 47.1 (12.94) | 58.2 (16.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 18 | 16 | 15 | 17 | 19 | 13 | 20 | 13 | 15 | 19 | 16 | 20 | 84 | 74 | 59 | 19 | 23 | 20 | 18 | 16 | 22 | 13 | 579
  Male | 15 | 13 | 12 | 14 | 15 | 15 | 14 | 19 | 13 | 20 | 18 | 14 | 13 | 12 | 40 | 48 | 55 | 12 | 7 | 13 | 12 | 10 | 10 | 16 | 430
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 22 | 22 | 23 | 24 | 26 | 3 | 8 | 9 | 7 | 9 | 15 | 18 | 18 | 47 | 42 | 47 | 11 | 8 | 10 | 9 | 8 | 12 | 9 | 432
  Not Hispanic or Latino | 5 | 6 | 8 | 7 | 6 | 6 | 27 | 24 | 24 | 24 | 24 | 18 | 11 | 14 | 77 | 79 | 67 | 20 | 22 | 23 | 21 | 18 | 20 | 20 | 571
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 11 | 8 | 5 | 2 | 2 | 2 | 4 | 3 | 2 | 3 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 1 | 5 | 1 | 3 | 5 | 1 | 1 | 0 | 5 | 2 | 1 | 3 | 8 | 12 | 6 | 12 | 0 | 5 | 6 | 7 | 7 | 5 | 3 | 103
  White | 24 | 27 | 24 | 29 | 25 | 27 | 32 | 30 | 33 | 26 | 30 | 32 | 24 | 23 | 100 | 104 | 95 | 28 | 22 | 24 | 19 | 14 | 25 | 22 | 839
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: SSA: Percentage of Participants With Local Reactions up to 7 Days Following Vaccination (18-64 Years)
Description: Local reactions included pain at the injection site, redness and swelling and were recorded by participants in an electronic diary. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 centimeter (cm). Redness and swelling were graded as mild (Grade 1): greater than (>) 2.0 cm to 5.0 cm; moderate (Grade 2): >5.0 cm to 10.0 cm; severe (Grade 3): >10 cm; potentially life-threatening (Grade 4): necrosis or exfoliative dermatitis (redness) and necrosis (swelling). Pain at injection site was graded as mild (Grade 1): did not interfere with activity; moderate (Grade 2): interfered with activity; severe (Grade 3): prevented daily activity and potentially life-threatening (Grade 4): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Percentage of participants with any local reactions were reported in this outcome measure.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32
Percentage of participants | 83.3 [65.3 to 94.4] | 89.3 [71.8 to 97.7] | 80.0 [61.4 to 92.3] | 63.3 [43.9 to 80.1] | 73.3 [54.1 to 87.7] | 71.9 [53.3 to 86.3]

2. Primary Outcome: SSA: Percentage of Participants With Local Reactions up to 7 Days Following Vaccination (>=65 Years)
Description: Local reactions included pain at the injection site, redness and swelling and were recorded by participants in an electronic diary. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 cm. Redness and swelling were graded as mild (Grade 1): >2.0 cm to 5.0 cm; moderate (Grade 2): >5.0 cm to 10.0 cm; severe (Grade 3): >10 cm; potentially life-threatening (Grade 4): necrosis or exfoliative dermatitis. Pain at injection site was graded as mild (Grade 1): did not interfere with activity; moderate (Grade 2): interfered with activity; severe (Grade 3): prevented daily activity and potentially life-threatening (Grade 4): emergency room visit or hospitalization for severe pain. Grade 4 reactions were classified by the investigator or medically qualified person. Percentage of participants with any local reactions were reported in this outcome measure.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 84.8 [68.1 to 94.9] | 53.1 [34.7 to 70.9] | 84.8 [68.1 to 94.9] | 63.6 [45.1 to 79.6] | 72.7 [54.5 to 86.7] | 51.5 [33.5 to 69.2]

3. Primary Outcome: SSA: Percentage of Participants With Systemic Events up to 7 Days Following Vaccination (18-64 Years)
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, chills, new or worsened muscle pain and new or worsened joint pain. Events were recorded by participants in an electronic diary. Fever defined as oral temperature >=38.0 deg C and categorized as>=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Vomiting graded as: G1: 1-2 times in 24 h; G2: >2 times in 24h; G3: required IV hydration. Diarrhea graded as: G1: 2-3 loose stools in 24h; G2: 4-5 loose stools in 24h; G3: 6 or more loose stools in 24h.Headache, fatigue, chills, new/worsened muscle pain and new/worsened joint pain: G1: didn't interfere with activity; G2: some interference with activity; G3: prevented daily routine activity. For all systemic events except fever, Grade 4=emergency room visit or hospitalization. Grade 4 events were classified by the investigator. Percentage of participants with any systemic events were reported in this outcome measure.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32
Percentage of participants | 76.7 [57.7 to 90.1] | 78.6 [59.0 to 91.7] | 70.0 [50.6 to 85.3] | 53.3 [34.3 to 71.7] | 63.3 [43.9 to 80.1] | 68.8 [50.0 to 83.9]

4. Primary Outcome: SSA: Percentage of Participants With Systemic Events up to 7 Days Following Vaccination (>=65 Years)
Description: as for outcome 3
Time Frame: SSA: From Day 1 to Day 7 after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 72.7 [54.5 to 86.7] | 50.0 [31.9 to 68.1] | 69.7 [51.3 to 84.4] | 45.5 [28.1 to 63.6] | 60.6 [42.1 to 77.1] | 45.5 [28.1 to 63.6]

5. Primary Outcome: SSA: Percentage of Participants Reporting AEs From Vaccination Through 4 Weeks After Vaccination (18-64 Years)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious AEs. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event. Only AEs collected by non-systematic assessment (excluding local reactions and systematic events) were included in this outcome measure.
Time Frame: SSA: From Vaccination on Day 1 through 4 Weeks after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32
Percentage of participants | 3.3 [0.1 to 17.2] | 10.7 [2.3 to 28.2] | 0 [0.0 to 11.6] | 3.3 [0.1 to 17.2] | 6.7 [0.8 to 22.1] | 3.1 [0.1 to 16.2]

6. Primary Outcome: SSA: Percentage of Participants Reporting Adverse Events From Vaccination Through 4 Weeks After Vaccination (>=65 Years)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs included both serious and all non-serious AEs. An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event. Only AEs collected by non-systematic assessment (excluding local reactions and systematic events) were included in this outcome measure.
Time Frame: SSA: From Vaccination on Day 1 through 4 Weeks after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 24.2 [11.1 to 42.3] | 9.4 [2.0 to 25.0] | 6.1 [0.7 to 20.2] | 6.1 [0.7 to 20.2] | 9.1 [1.9 to 24.3] | 0 [0.0 to 10.6]

7. Primary Outcome: SSA: Percentage of Participants Reporting Serious Adverse Events (SAEs) From Vaccination Through 6 Months After Vaccination (18-64 Years)
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event.
Time Frame: SSA: From Vaccination on Day 1 through 6 Months after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32
Percentage of participants | 0 [0.0 to 11.6] | 3.6 [0.1 to 18.3] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 3.1 [0.1 to 16.2]

8. Primary Outcome: SSA: Percentage of Participants Reporting SAEs From Vaccination Through 6 Months After Vaccination (>=65 Years)
Description: as for outcome 7
Time Frame: SSA: From Vaccination on Day 1 through 6 Months after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 0 [0.0 to 10.6] | 0 [0.0 to 10.9] | 0 [0.0 to 10.6] | 6.1 [0.7 to 20.2] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6]

9. Primary Outcome: SSA: Percentage of Participants With Abnormal Serum Troponin 1 Laboratory Values at 2 Days After Vaccination (18-64 Years)
Description: An abnormal troponin 1 result was defined as any troponin 1 level >=0.30 nanogram per milliliter.
Time Frame: SSA: 2 Days after Vaccination
Population: Safety population included all participants who received the study intervention. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Participants were analyzed according to the treatment which they received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 28 | 28 | 29 | 29 | 30
Percentage of participants | 0 [0.0 to 12.3] | 0 [0.0 to 12.3] | 0 [0.0 to 12.3] | 0 [0.0 to 11.9] | 0 [0.0 to 11.9] | 0 [0.0 to 11.6]

10. Primary Outcome: SSA: Percentage of Participants With Abnormal Serum Troponin 1 Laboratory Values at 2 Days After Vaccination (>=65 Years)
Description: An abnormal troponin 1 result was defined as any troponin 1 level >=0.30 nanogram per milliliter.
Time Frame: SSA: 2 Days after Vaccination
Population: Safety population included all participants who received the study intervention. Here, "Number of Participants Analyzed" signifies participants evaluable for this outcome measure. Participants were analyzed according to the treatment to which they were received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 30 | 31 | 32 | 31 | 32
Percentage of participants | 0 [0.0 to 10.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 11.2] | 0 [0.0 to 10.9]

11. Primary Outcome: SSA: Percentage of Participants With Abnormal Serum Troponin 1 Laboratory Values at 1 Week After Vaccination (18-64 Years)
Description: An abnormal troponin 1 result was defined as any troponin 1 level >=0.30 nanogram per milliliter.
Time Frame: SSA: 1 Week After Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 26 | 29 | 30 | 30 | 31
Percentage of participants | 3.3 [0.1 to 17.2] | 0 [0.0 to 13.2] | 0 [0.0 to 11.9] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2]

12. Primary Outcome: SSA: Percentage of Participants With Abnormal Serum Troponin 1 Laboratory Values at 1 Week After Vaccination (>=65 Years)
Description: An abnormal troponin 1 result was defined as any troponin 1 level >=0.30 nanogram per milliliter.
Time Frame: SSA: 1 Week After Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 31 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6]

13. Primary Outcome: SSA: Percentage of Participants With New Electrocardiogram (ECG) Abnormalities at 2 Days After Vaccination (18-64 Years)
Description: An ECG abnormality was defined as any new abnormality that, as judged by a cardiologist, was consistent with probable or possible myocarditis or pericarditis, including: sustained atrial or ventricular arrhythmias, second-degree Mobitz Type II or worse atrioventricular block, new bundle branch block and diffuse ST-segment elevation or PR-segment inversion, compatible with pericarditis.
Time Frame: SSA: 2 Days after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32
Percentage of participants | 0 [0.0 to 11.6] | 0 [0.0 to 12.3] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9]

14. Primary Outcome: SSA: Percentage of Participants With New ECG Abnormalities at 2 Days After Vaccination (>=65 Years)
Description: as for outcome 13
Time Frame: SSA: 2 Days after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 0 [0.0 to 10.6] | 0 [0.0 to 10.9] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6]

15. Primary Outcome: SSA: Percentage of Participants With New ECG Abnormalities at 1 Week After Vaccination (18-64 Years)
Description: as for outcome 13
Time Frame: SSA: 1 Week after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 30 | 28 | 30 | 30 | 30 | 32
Percentage of participants | 0 [0.0 to 11.6] | 0 [0.0 to 12.3] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 10.9]

16. Primary Outcome: SSA: Percentage of Participants With New ECG Abnormalities at 1 Week After Vaccination (>=65 Years)
Description: as for outcome 13
Time Frame: SSA: 1 Week after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 33 | 32 | 33 | 33 | 33 | 33
Percentage of participants | 0 [0.0 to 10.6] | 0 [0.0 to 10.9] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6] | 0 [0.0 to 10.6]

17. Primary Outcome: SSB: Percentage of Participants With Abnormal Serum Troponin 1 Laboratory Values at 2 Days After Vaccination (18- 64 Years)
Description: An abnormal troponin 1 result was defined as any troponin 1 level >=0.30 nanogram per milliliter.
Time Frame: SSB: 2 Days after Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 31 | 123 | 122 | 113 | 31 | 29 | 32 | 29 | 26 | 32 | 28
Percentage of participants | 0 [0.0 to 11.9] | 0 [0.0 to 11.2] | 0 [0.0 to 3.0] | 0 [0.0 to 3.0] | 0 [0.0 to 3.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9] | 0 [0.0 to 13.2] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3]

18. Primary Outcome: SSB: Percentage of Participants With Abnormal Serum Troponin 1 Laboratory Values at 1 Week After Vaccination (18- 64 Years)
Description: An abnormal troponin 1 result was defined as any troponin 1 level >=0.30 nanogram per milliliter.
Time Frame: SSB: 1 Week after Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 121 | 120 | 111 | 30 | 30 | 33 | 30 | 26 | 32 | 28
Percentage of participants | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [0.0 to 3.0] | 0 [0.0 to 3.0] | 0 [0.0 to 3.3] | 0 [0.0 to 11.6] | 0 [0.0 to 11.6] | 0 [0.0 to 10.6] | 0 [0.0 to 11.6] | 0 [0.0 to 13.2] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3]

19. Primary Outcome: SSB: Percentage of Participants With New ECG Abnormalities at 2 Days After Vaccination (18- 64 Years)
Description: as for outcome 13
Time Frame: SSB: 2 Days after Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 123 | 122 | 113 | 31 | 30 | 33 | 30 | 26 | 32 | 28
Percentage of participants | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [0.0 to 3.0] | 0 [0.0 to 3.0] | 0 [0.0 to 3.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.6] | 0 [0.0 to 11.6] | 0 [0.0 to 13.2] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3]

20. Primary Outcome: SSB: Percentage of Participants With New ECG Abnormalities at 1 Week After Vaccination (18- 64 Years)
Description: as for outcome 13
Time Frame: SSB: 1 Week after Vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 123 | 122 | 113 | 31 | 30 | 33 | 30 | 26 | 32 | 28
Percentage of participants | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [0.0 to 3.0] | 0 [0.0 to 3.0] | 0 [0.0 to 3.2] | 0 [0.0 to 11.2] | 0 [0.0 to 11.6] | 0 [0.0 to 10.6] | 0 [0.0 to 11.6] | 0 [0.0 to 13.2] | 0 [0.0 to 10.9] | 0 [0.0 to 12.3]

21. Primary Outcome: SSB: Percentage of Participants With Local Reactions up to 7 Days Following Vaccination (18- 64 Years)
Description: as for outcome 2
Time Frame: SSB: From Day 1 to Day 7 after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 124 | 122 | 114 | 31 | 30 | 33 | 30 | 26 | 32 | 29
Percentage of participants | 58.6 [38.9 to 76.5] | 71.9 [53.3 to 86.3] | 78.2 [69.9 to 85.1] | 82.8 [74.9 to 89.0] | 75.4 [66.5 to 83.0] | 80.6 [62.5 to 92.5] | 80.0 [61.4 to 92.3] | 81.8 [64.5 to 93.0] | 66.7 [47.2 to 82.7] | 73.1 [52.2 to 88.4] | 71.9 [53.3 to 86.3] | 69.0 [49.2 to 84.7]

22. Primary Outcome: SSB: Percentage of Participants With Systemic Events up to 7 Days Following Vaccination (18- 64 Years)
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, chills, new or worsened muscle pain and new or worsened joint pain. Events were recorded by participants in an electronic diary. Fever defined as oral temperature >=38.0 deg C and categorized as >=38.0 to 38.4 deg C, >38.4 to 38.9 deg C, >38.9 to 40.0 deg C and >40.0 deg C. Vomiting graded as: G1: 1-2 times in 24 h; G2: >2 times in 24h; G3: required IV hydration. Diarrhea graded as: G1: 2-3 loose stools in 24h; G2: 4-5 loose stools in 24h; G3: 6 or more loose stools in 24h. Headache, fatigue, chills, new/worsened muscle pain and new/worsened joint pain: G1: didn't interfere with activity; G2: some interference with activity; G3: prevented daily routine activity. For all systemic events except fever, Grade 4=emergency room visit or hospitalization. Grade 4 events were classified by the investigator. Percentage of participants with any systemic events were reported in this outcome measure.
Time Frame: SSB: From Day 1 to Day 7 after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 124 | 122 | 114 | 31 | 30 | 33 | 30 | 26 | 32 | 29
Percentage of participants | 51.7 [32.5 to 70.6] | 62.5 [43.7 to 78.9] | 74.2 [65.6 to 81.6] | 77.0 [68.6 to 84.2] | 71.1 [61.8 to 79.2] | 80.6 [62.5 to 92.5] | 80.0 [61.4 to 92.3] | 72.7 [54.5 to 86.7] | 73.3 [54.1 to 87.7] | 65.4 [44.3 to 82.8] | 68.8 [50.0 to 83.9] | 48.3 [29.4 to 67.5]

23. Primary Outcome: SSB: Percentage of Participants Reporting AEs From Vaccination Through 4 Weeks After Vaccination (18- 64 Years)
Description: as for outcome 6
Time Frame: SSB: From Vaccination on Day 1 through 4 Weeks after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 124 | 122 | 114 | 31 | 30 | 33 | 30 | 26 | 32 | 29
Percentage of participants | 0 [0.0 to 11.9] | 3.1 [0.1 to 16.2] | 4.8 [1.8 to 10.2] | 6.6 [2.9 to 12.5] | 6.1 [2.5 to 12.2] | 9.7 [2.0 to 25.8] | 6.7 [0.8 to 22.1] | 6.1 [0.7 to 20.2] | 6.7 [0.8 to 22.1] | 0 [0.0 to 13.2] | 9.4 [2.0 to 25.0] | 0 [0.0 to 11.9]

24. Primary Outcome: SSB: Percentage of Participants Reporting SAEs From Vaccination Through 6 Months After Vaccination (18- 64 Years)
Description: as for outcome 7
Time Frame: SSB: From Vaccination on Day 1 through 6 Months after Vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 29 | 32 | 124 | 122 | 114 | 31 | 30 | 33 | 30 | 26 | 32 | 29
Percentage of participants | 0 [0.0 to 11.9] | 0 [0.0 to 10.9] | 0 [0.0 to 2.9] | 0 [0.0 to 3.0] | 0 [0.0 to 3.2] | 3.2 [0.1 to 16.7] | 0 [0.0 to 11.6] | 0 [0.0 to 10.6] | 0 [0.0 to 11.6] | 0 [0.0 to 13.2] | 0 [0.0 to 10.9] | 0 [0.0 to 11.9]

25. Secondary Outcome: SSA: Geometric Mean Titers (GMTs) of Strain-Specific Hemagglutination Inhibition (HAI) Before Vaccination and at 4 Weeks After Vaccination (18- 64 Years)
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria and B/Phuket.
Time Frame: SSA: Before Vaccination and 4 Weeks after Vaccination
Population: Evaluable immunogenicity population (EIP) included all eligible participants who receive the study intervention to which they were randomized; had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 30 | 28 | 31
Titers
  A/Wisconsin: Before vaccination: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  A/Wisconsin: Before vaccination | 32.0 [16.6 to 61.8] | 14.7 [8.8 to 24.7] | 31.2 [18.4 to 53.0] | 26.0 [16.6 to 40.7] | 16.4 [9.5 to 28.2] | 34.2 [19.5 to 59.9]
  A/Wisconsin: 4 Weeks after vaccination | 341.6 [226.5 to 515.4] | 201.6 [121.0 to 335.8] | 282.7 [164.3 to 486.5] | 259.9 [177.9 to 379.8] | 249.8 [153.6 to 406.3] | 294.7 [184.9 to 469.9]
  A/Darwin: Before vaccination: number analyzed (Participants) | 28 | 25 | 27 | 29 | 28 | 31
  A/Darwin: Before vaccination | 32.0 [18.9 to 54.3] | 31.2 [18.5 to 52.5] | 30.9 [20.1 to 47.6] | 23.6 [15.0 to 37.3] | 16.4 [10.1 to 26.8] | 36.6 [25.6 to 52.3]
  A/Darwin: 4 Weeks after vaccination: number analyzed (Participants) | 27 | 27 | 28 | 30 | 28 | 31
  A/Darwin: 4 Weeks after vaccination | 165.5 [101.0 to 271.2] | 141.9 [83.1 to 242.2] | 160.0 [102.5 to 249.7] | 167.6 [120.2 to 233.7] | 129.1 [77.9 to 213.7] | 97.8 [62.9 to 152.1]
  B/Austria: Before vaccination: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  B/Austria: Before vaccination | 10.5 [7.0 to 15.8] | 12.0 [7.4 to 19.3] | 11.0 [7.2 to 16.9] | 9.8 [6.7 to 14.1] | 10.5 [7.1 to 15.6] | 12.0 [7.9 to 18.0]
  B/Austria: 4 Weeks after vaccination | 14.9 [9.5 to 23.2] | 20.0 [12.4 to 32.4] | 18.6 [11.7 to 29.4] | 17.8 [11.2 to 28.3] | 20.0 [12.0 to 33.2] | 40.0 [24.8 to 64.5]
  B/Phuket: Before vaccination: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  B/Phuket: Before vaccination | 18.1 [12.0 to 27.3] | 16.7 [10.5 to 26.5] | 12.8 [8.5 to 19.4] | 21.0 [13.3 to 33.1] | 12.2 [8.6 to 17.3] | 24.5 [16.2 to 36.9]
  B/Phuket: 4 Weeks after vaccination | 26.9 [17.3 to 41.9] | 36.1 [24.2 to 53.9] | 35.3 [22.6 to 55.2] | 45.9 [30.0 to 70.4] | 41.0 [27.9 to 60.2] | 78.2 [55.5 to 110.4]

26. Secondary Outcome: SSA: GMTs of Strain-Specific HAI Before Vaccination and at 4 Weeks After Vaccination (>=65 Years)
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria and B/Phuket.
Time Frame: SSA: Before Vaccination and 4 Weeks after Vaccination
Population: EIP included all eligible participants who receive the study intervention to which they were randomized; had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 29 | 32
Titers
  A/Wisconsin: Before vaccination | 56.6 [35.5 to 90.2] | 38.3 [24.3 to 60.3] | 57.8 [36.1 to 92.6] | 53.5 [36.1 to 79.2] | 69.3 [45.1 to 106.6] | 50.8 [34.2 to 75.3]
  A/Wisconsin: 4 Weeks after vaccination | 113.1 [73.9 to 173.2] | 97.2 [69.0 to 137.0] | 156.6 [97.6 to 251.2] | 119.6 [82.6 to 173.2] | 150.1 [95.2 to 236.6] | 80.0 [56.8 to 112.6]
  A/Darwin: Before vaccination: number analyzed (Participants) | 31 | 32 | 30 | 31 | 29 | 32
  A/Darwin: Before vaccination | 57.2 [38.6 to 84.8] | 40.9 [31.3 to 53.3] | 62.0 [46.7 to 82.4] | 41.8 [29.6 to 59.2] | 71.0 [52.2 to 96.6] | 56.6 [37.3 to 85.8]
  A/Darwin: 4 Weeks after vaccination | 107.5 [75.4 to 153.3] | 115.6 [84.7 to 157.8] | 134.5 [96.2 to 188.3] | 81.8 [61.2 to 109.3] | 181.7 [120.5 to 274.1] | 83.5 [57.4 to 121.6]
  B/Austria: Before vaccination | 37.5 [26.9 to 52.2] | 28.3 [17.4 to 45.9] | 27.1 [18.8 to 39.0] | 28.0 [18.2 to 43.0] | 44.0 [28.9 to 67.1] | 22.8 [16.5 to 31.4]
  B/Austria: 4 Weeks after vaccination | 49.7 [37.8 to 65.2] | 44.6 [28.8 to 68.9] | 40.9 [29.3 to 57.0] | 40.9 [28.6 to 58.4] | 64.5 [44.7 to 93.1] | 41.8 [32.7 to 53.4]
  B/Phuket: Before vaccination | 14.8 [10.8 to 20.3] | 11.9 [8.9 to 15.9] | 12.4 [8.7 to 17.6] | 10.7 [8.0 to 14.3] | 15.0 [10.6 to 21.3] | 10.4 [7.9 to 13.8]
  B/Phuket: 4 Weeks after vaccination | 20.0 [15.1 to 26.6] | 14.5 [10.8 to 19.3] | 20.4 [14.2 to 29.5] | 15.0 [11.1 to 20.2] | 26.0 [18.0 to 37.6] | 15.4 [11.0 to 21.7]

27. Secondary Outcome: SSA: Geometric Mean Fold Rise (GMFRs) of Strain-Specific HAI From Before Vaccination to 4 Weeks After Vaccination (18- 64 Years)
Description: GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. When pre-vaccination assay results were lower than the LLOQ and the post-vaccination results were greater than or equal to the LLOQ, the pre-vaccination assay results were set to LLOQ for the GMFR calculation. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria and B/Phuket.
Time Frame: SSA: Before Vaccination to 4 Weeks after Vaccination
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 30 | 28 | 31
Fold Rise
  A/Wisconsin: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  A/Wisconsin | 8.5 [4.8 to 15.2] | 9.8 [5.7 to 16.8] | 8.2 [3.9 to 17.2] | 9.7 [5.9 to 15.9] | 11.0 [6.7 to 18.1] | 7.5 [4.1 to 13.9]
  A/Darwin: number analyzed (Participants) | 27 | 25 | 27 | 29 | 28 | 31
  A/Darwin | 4.1 [2.7 to 6.3] | 3.9 [2.5 to 6.1] | 4.7 [3.0 to 7.3] | 5.9 [3.9 to 8.8] | 5.7 [3.8 to 8.6] | 2.5 [1.7 to 3.7]
  B/Austria: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  B/Austria | 1.2 [0.9 to 1.6] | 1.3 [1.1 to 1.7] | 1.4 [1.0 to 1.9] | 1.7 [1.2 to 2.3] | 1.6 [1.1 to 2.2] | 2.6 [1.7 to 3.9]
  B/Phuket: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  B/Phuket | 1.3 [1.0 to 1.8] | 1.8 [1.4 to 2.4] | 2.2 [1.6 to 3.1] | 1.9 [1.5 to 2.5] | 2.6 [1.9 to 3.6] | 2.7 [2.0 to 3.7]

28. Secondary Outcome: SSA: GMFRs of Strain-Specific HAI From Before Vaccination to 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 27
Time Frame: SSA: Before Vaccination to 4 Weeks after Vaccination
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 29 | 32
Fold Rise
  A/Wisconsin | 2.0 [1.6 to 2.4] | 2.3 [1.8 to 3.0] | 2.7 [2.1 to 3.4] | 2.2 [1.7 to 2.9] | 2.2 [1.7 to 2.7] | 1.5 [1.1 to 2.2]
  A/Darwin: number analyzed (Participants) | 31 | 32 | 30 | 31 | 29 | 32
  A/Darwin | 1.8 [1.5 to 2.2] | 2.8 [2.1 to 3.7] | 2.1 [1.7 to 2.7] | 1.9 [1.5 to 2.3] | 2.6 [1.9 to 3.5] | 1.4 [1.0 to 2.0]
  B/Austria | 1.3 [1.1 to 1.6] | 1.4 [1.2 to 1.7] | 1.4 [1.2 to 1.7] | 1.3 [1.1 to 1.6] | 1.4 [1.1 to 1.8] | 1.7 [1.3 to 2.2]
  B/Phuket | 1.2 [1.1 to 1.4] | 1.1 [1.0 to 1.3] | 1.4 [1.1 to 1.6] | 1.2 [1.1 to 1.4] | 1.5 [1.2 to 1.9] | 1.4 [1.1 to 1.7]

29. Secondary Outcome: SSA: Percentage of Participants Achieving HAI Seroconversion for Each Strain at 4 Weeks After Vaccination (18- 64 Years)
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria and B/Phuket.
Time Frame: SSA: 4 Weeks after Vaccination
Population: EIP included all eligible participants who receive study intervention to which they were randomized;had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations."Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
Percentage of participants
  A/Wisconsin | 75.0 [55.1 to 89.3] | 77.8 [57.7 to 91.4] | 71.4 [51.3 to 86.8] | 86.2 [68.3 to 96.1] | 89.3 [71.8 to 97.7] | 61.3 [42.2 to 78.2]
  A/Darwin: number analyzed (Participants) | 27 | 25 | 27 | 29 | 28 | 31
  A/Darwin | 63.0 [42.4 to 80.6] | 60.0 [38.7 to 78.9] | 70.4 [49.8 to 86.2] | 69.0 [49.2 to 84.7] | 75.0 [55.1 to 89.3] | 35.5 [19.2 to 54.6]
  B/Austria | 14.3 [4.0 to 32.7] | 3.7 [0.1 to 19.0] | 21.4 [8.3 to 41.0] | 17.2 [5.8 to 35.8] | 25.0 [10.7 to 44.9] | 38.7 [21.8 to 57.8]
  B/Phuket | 17.9 [6.1 to 36.9] | 18.5 [6.3 to 38.1] | 32.1 [15.9 to 52.4] | 34.5 [17.9 to 54.3] | 50.0 [30.6 to 69.4] | 38.7 [21.8 to 57.8]

30. Secondary Outcome: SSA: Percentage of Participants Achieving HAI Seroconversion for Each Strain at 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 29
Time Frame: SSA: 4 Weeks after Vaccination
Population: EIP included all eligible participants who receive study intervention to which they were randomized;had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 29 | 32
Percentage of participants
  A/Wisconsin | 15.6 [5.3 to 32.8] | 25.0 [11.5 to 43.4] | 46.9 [29.1 to 65.3] | 32.3 [16.7 to 51.4] | 34.5 [17.9 to 54.3] | 12.5 [3.5 to 29.0]
  A/Darwin: number analyzed (Participants) | 31 | 32 | 30 | 31 | 29 | 32
  A/Darwin | 12.9 [3.6 to 29.8] | 43.8 [26.4 to 62.3] | 30.0 [14.7 to 49.4] | 19.4 [7.5 to 37.5] | 41.4 [23.5 to 61.1] | 12.5 [3.5 to 29.0]
  B/Austria | 9.4 [2.0 to 25.0] | 6.3 [0.8 to 20.8] | 6.3 [0.8 to 20.8] | 6.5 [0.8 to 21.4] | 6.9 [0.8 to 22.8] | 15.6 [5.3 to 32.8]
  B/Phuket | 0 [0.0 to 10.9] | 3.1 [0.1 to 16.2] | 9.4 [2.0 to 25.0] | 0 [0.0 to 11.2] | 13.8 [3.9 to 31.7] | 12.5 [3.5 to 29.0]

31. Secondary Outcome: SSA: Percentage of Participants With Strain Specific HAI Titers Greater Than or Equal to (>=) 1:40 Before Vaccination and at 4 Weeks After Vaccination (18- 64 Years)
Description: Percentage of participants with HAI titer >=1:40 for each strain before vaccination and 4 weeks after vaccination is presented in this outcome measure. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria and B/Phuket.
Time Frame: SSA: Before Vaccination and at 4 Weeks after Vaccination
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 30 | 28 | 31
Percentage of participants
  A/Wisconsin: Before Vaccination: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  A/Wisconsin: Before Vaccination | 53.6 [33.9 to 72.5] | 25.9 [11.1 to 46.3] | 46.4 [27.5 to 66.1] | 44.8 [26.4 to 64.3] | 32.1 [15.9 to 52.4] | 58.1 [39.1 to 75.5]
  A/Wisconsin: 4 Weeks After Vaccination | 96.4 [81.7 to 99.9] | 92.6 [75.7 to 99.1] | 92.9 [76.5 to 99.1] | 96.7 [82.8 to 99.9] | 100.0 [87.7 to 100.0] | 96.8 [83.3 to 99.9]
  A/Darwin: Before Vaccination: number analyzed (Participants) | 28 | 25 | 27 | 29 | 28 | 31
  A/Darwin: Before Vaccination | 60.7 [40.6 to 78.5] | 56.0 [34.9 to 75.6] | 66.7 [46.0 to 83.5] | 51.7 [32.5 to 70.6] | 42.9 [24.5 to 62.8] | 67.7 [48.6 to 83.3]
  A/Darwin: 4 Weeks After Vaccination: number analyzed (Participants) | 27 | 27 | 28 | 30 | 28 | 31
  A/Darwin: 4 Weeks After Vaccination | 85.2 [66.3 to 95.8] | 92.6 [75.7 to 99.1] | 96.4 [81.7 to 99.9] | 96.7 [82.8 to 99.9] | 85.7 [67.3 to 96.0] | 87.1 [70.2 to 96.4]
  B/Austria: Before Vaccination: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  B/Austria: Before Vaccination | 14.3 [4.0 to 32.7] | 25.9 [11.1 to 46.3] | 17.9 [6.1 to 36.9] | 13.8 [3.9 to 31.7] | 21.4 [8.3 to 41.0] | 22.6 [9.6 to 41.1]
  B/Austria: 4 Weeks After Vaccination | 28.6 [13.2 to 48.7] | 33.3 [16.5 to 54.0] | 42.9 [24.5 to 62.8] | 33.3 [17.3 to 52.8] | 39.3 [21.5 to 59.4] | 54.8 [36.0 to 72.7]
  B/Phuket: Before Vaccination: number analyzed (Participants) | 28 | 27 | 28 | 29 | 28 | 31
  B/Phuket: Before Vaccination | 32.1 [15.9 to 52.4] | 25.9 [11.1 to 46.3] | 14.3 [4.0 to 32.7] | 48.3 [29.4 to 67.5] | 21.4 [8.3 to 41.0] | 51.6 [33.1 to 69.8]
  B/Phuket: 4 Weeks After Vaccination | 57.1 [37.2 to 75.5] | 55.6 [35.3 to 74.5] | 53.6 [33.9 to 72.5] | 70.0 [50.6 to 85.3] | 67.9 [47.6 to 84.1] | 90.3 [74.2 to 98.0]

32. Secondary Outcome: SSA: Percentage of Participants With Strain Specific HAI Titers >= 1:40 Before Vaccination and at 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 31
Time Frame: SSA: Before Vaccination and at 4 Weeks After Vaccination
Population: as for outcome 26
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 29 | 32
Percentage of participants
  A/Wisconsin: Before Vaccination | 68.8 [50.0 to 83.9] | 59.4 [40.6 to 76.3] | 62.5 [43.7 to 78.9] | 71.0 [52.0 to 85.8] | 75.9 [56.5 to 89.7] | 75.0 [56.6 to 88.5]
  A/Wisconsin: 4 Weeks After Vaccination | 90.6 [75.0 to 98.0] | 96.9 [83.8 to 99.9] | 87.5 [71.0 to 96.5] | 93.5 [78.6 to 99.2] | 93.1 [77.2 to 99.2] | 93.8 [79.2 to 99.2]
  A/Darwin: Before Vaccination: number analyzed (Participants) | 31 | 32 | 30 | 31 | 29 | 32
  A/Darwin: Before Vaccination | 83.9 [66.3 to 94.5] | 81.3 [63.6 to 92.8] | 86.7 [69.3 to 96.2] | 74.2 [55.4 to 88.1] | 89.7 [72.6 to 97.8] | 78.1 [60.0 to 90.7]
  A/Darwin: 4 Weeks After Vaccination | 93.8 [79.2 to 99.2] | 100.0 [89.1 to 100.0] | 96.9 [83.8 to 99.9] | 87.1 [70.2 to 96.4] | 100.0 [88.1 to 100.0] | 90.6 [75.0 to 98.0]
  B/Austria: Before Vaccination | 62.5 [43.7 to 78.9] | 56.3 [37.7 to 73.6] | 53.1 [34.7 to 70.9] | 54.8 [36.0 to 72.7] | 62.1 [42.3 to 79.3] | 43.8 [26.4 to 62.3]
  B/Austria: 4 Weeks After Vaccination | 75.0 [56.6 to 88.5] | 62.5 [43.7 to 78.9] | 65.6 [46.8 to 81.4] | 64.5 [45.4 to 80.8] | 75.9 [56.5 to 89.7] | 68.8 [50.0 to 83.9]
  B/Phuket: Before Vaccination | 25.0 [11.5 to 43.4] | 15.6 [5.3 to 32.8] | 15.6 [5.3 to 32.8] | 9.7 [2.0 to 25.8] | 31.0 [15.3 to 50.8] | 12.5 [3.5 to 29.0]
  B/Phuket: 4 Weeks After Vaccination | 31.3 [16.1 to 50.0] | 21.9 [9.3 to 40.0] | 31.3 [16.1 to 50.0] | 25.8 [11.9 to 44.6] | 51.7 [32.5 to 70.6] | 31.3 [16.1 to 50.0]

33. Secondary Outcome: SSA: Percentage of Participants Achieving HAI Seroconversion for All Strains at 4 Weeks After Vaccination (18- 64 Years)
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Data is reported combined for all strains (A/Wisconsin, A/Darwin, B/Austria and B/Phuket).
Time Frame: SSA: 4 Weeks after Vaccination
Population: EIP included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations before vaccination. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 27 | 25 | 27 | 29 | 28 | 31
Percentage of participants | 3.7 [0.1 to 19.0] | 0 [0.0 to 13.7] | 7.4 [0.9 to 24.3] | 3.4 [0.1 to 17.8] | 10.7 [2.3 to 28.2] | 6.5 [0.8 to 21.4]

34. Secondary Outcome: SSA: Percentage of Participants Achieving HAI Seroconversion for All Strains at 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 33
Time Frame: SSA: 4 Weeks after Vaccination
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 31 | 32 | 30 | 31 | 29 | 32
Percentage of participants | 0 [0.0 to 11.2] | 0 [0.0 to 10.9] | 0 [0.0 to 11.6] | 0 [0.0 to 11.2] | 3.4 [0.1 to 17.8] | 3.1 [0.1 to 16.2]

35. Secondary Outcome: SSA: Percentage of Participants With HAI Titers >= 1.40 for All Strain at 4 Weeks After Vaccination (18- 64 Years)
Description: Percentage of participants achieving HAI titers >= 1:40 for each strain at 4 weeks after last vaccination is reported in this outcome measure. Exact 2-sided CI was based on the Clopper and Pearson method. Data is reported combined for all strains (A/Wisconsin, A/Darwin, B/Austria and B/Phuket).
Time Frame: SSA: 4 Weeks after Vaccination
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 27 | 27 | 28 | 30 | 28 | 31
Percentage of participants | 18.5 [6.3 to 38.1] | 22.2 [8.6 to 42.3] | 21.4 [8.3 to 41.0] | 26.7 [12.3 to 45.9] | 28.6 [13.2 to 48.7] | 51.6 [33.1 to 69.8]

36. Secondary Outcome: SSA: Percentage of Participants With HAI Titers >= 1.40 for All Strain at 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 35
Time Frame: SSA: 4 Weeks after Vaccination
Population: EIP included all eligible participants who receive the study intervention to which they were randomized; had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 31 | 29 | 32
Percentage of participants | 21.9 [9.3 to 40.0] | 15.6 [5.3 to 32.8] | 28.1 [13.7 to 46.7] | 22.6 [9.6 to 41.1] | 41.4 [23.5 to 61.1] | 21.9 [9.3 to 40.0]

37. Secondary Outcome: SSA: GMTs of SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers Before Vaccination and at 4 Weeks After Vaccination (18- 64 Years)
Description: GMT of SARS-CoV-2 Omicron (BA.4/BA.5)- neutralizing titers and SARS-CoV-2 reference strain (BNT162b2 Original [ancestral strain: Wuhan-Hu-1; USA-WA1/2020]) neutralizing titers before study vaccination and at 4 week after vaccination were reported in this outcome measure. GMT and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: SSA: Before Vaccination and 4 Weeks after Vaccination
Population: EIP included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations before vaccination. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Only arms which received covid vaccine (BNT162b2) were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 31
Titers
  SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers: Before Vaccination | 499.0 [298.2 to 835.0] | 240.9 [134.6 to 431.3] | 466.9 [277.8 to 784.7] | 415.8 [252.0 to 686.1]
  SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers: 4 Weeks After Vaccination | 3676.8 [2660.6 to 5081.2] | 2202.4 [1475.1 to 3288.4] | 2139.4 [1483.5 to 3085.3] | 3890.4 [2424.0 to 6243.6]
  SARS-CoV-2-Reference-Strain Neutralizing Titers: Before Vaccination | 3068.0 [2056.4 to 4577.1] | 1466.1 [869.2 to 2473.0] | 2487.1 [1541.8 to 4012.0] | 2719.1 [1828.8 to 4042.7]
  SARS-CoV-2-Reference-Strain Neutralizing Titers: 4 Weeks After Vaccination | 12713.5 [9538.2 to 16945.9] | 8069.0 [5808.1 to 11209.9] | 7166.0 [5568.6 to 9221.6] | 10719.9 [7287.6 to 15768.6]

38. Secondary Outcome: SSA: GMTs of SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers Before Vaccination and at 4 Weeks After Vaccination (>=65 Years)
Description: GMT of SARS-CoV-2 Omicron (BA.4/BA.5)- neutralizing titers and SARS-CoV-2 reference strain (BNT162b2 Original [ancestral strain: Wuhan-Hu-1; USA-WA1/2020]) neutralizing titers before study vaccination and at 4 week after vaccination was reported in this outcome measure. GMT and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the titers and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: SSA: Before Vaccination and 4 Weeks after Vaccination
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 32
Titers
  Omicron (BA.4/BA.5)- Neutralizing Titers: Before Vaccination | 1233.2 [635.1 to 2394.5] | 678.7 [347.6 to 1325.1] | 866.0 [434.5 to 1726.0] | 1472.6 [742.6 to 2920.3]
  Omicron (BA.4/BA.5)- Neutralizing Titers: 4 Weeks After Vaccination | 3627.4 [2167.0 to 6071.8] | 1841.1 [1113.0 to 3045.6] | 2770.7 [1483.7 to 5174.3] | 3774.4 [2434.8 to 5851.2]
  Reference-Strain Neutralizing Titers: Before Vaccination | 6045.7 [3580.2 to 10209.0] | 4567.0 [2725.1 to 7654.1] | 4461.1 [2766.5 to 7193.9] | 7654.1 [5009.9 to 11693.9]
  Reference-Strain Neutralizing Titers: 4 Weeks After Vaccination | 15305.0 [10000.4 to 23423.4] | 7821.2 [5348.8 to 11436.4] | 10280.2 [6847.9 to 15432.9] | 15646.0 [11782.3 to 20776.7]

39. Secondary Outcome: SSA: GMFR of SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers Before Vaccination to 4 Weeks After Vaccination (18- 64 Years)
Description: GMFR of SARS-CoV-2 Omicron (BA.4/BA.5)- neutralizing titers and SARS-CoV-2 reference strain (BNT162b2 Original [ancestral strain: Wuhan-Hu-1; USA-WA1/2020]) neutralizing titers before study vaccination to 4 week after vaccination was reported in this outcome measure. GMFR and the corresponding 2-sided CIs were calculated by exponentiating the mean logarithm of the fold rise and the corresponding CIs (based on Student's t distribution). Assay results below the LLOQ were set to 0.5*LLOQ.
Time Frame: SSA: Before Vaccination to 4 Weeks after Vaccination
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 31
Fold Rise
  Omicron (BA.4/BA.5)- Neutralizing Titers | 7.0 [4.7 to 10.4] | 7.6 [5.8 to 10.0] | 4.4 [2.7 to 7.1] | 8.7 [5.6 to 13.7]
  Reference-Strain Neutralizing Titers | 4.1 [3.0 to 5.8] | 5.5 [3.8 to 7.9] | 2.9 [1.9 to 4.5] | 3.9 [2.8 to 5.5]

40. Secondary Outcome: SSA: GMFR of SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers Before Vaccination to 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 39
Time Frame: SSA: Before Vaccination to 4 Weeks after Vaccination
Population: as for outcome 37
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 32
Fold Rise
  Omicron (BA.4/BA.5)- Neutralizing Titers | 2.8 [2.0 to 3.9] | 2.4 [1.8 to 3.3] | 3.0 [2.2 to 4.2] | 2.4 [1.7 to 3.4]
  Reference-Strain Neutralizing Titers | 2.5 [1.9 to 3.4] | 1.7 [1.3 to 2.3] | 2.3 [1.8 to 3.0] | 2.0 [1.5 to 2.7]

41. Secondary Outcome: SSA: Percentage of Participants With Seroresponse Based on SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers at 4 Weeks After Vaccination (18- 64 Years)
Description: Seroresponse was defined as achieving >= 4-fold rise from baseline (before study vaccination). If the baseline measurement was below the LLOQ, the postvaccination assay result of >= 4*LLOQ was considered a seroresponse. Exact 2-sided 95% CI, based on the Clopper and Pearson method. Percentage of participants achieving seroresponse Based on SARS-CoV-2 Omicron (BA.4/BA.5)- neutralizing titers and SARS-CoV-2-Reference-Strain (ancestral strain (Wuhan-Hu-1; USA-WA1/2020) neutralizing titers at 4 weeks after study vaccination was reported in this outcome measure.
Time Frame: SSA: 4 Weeks after Vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 28 | 27 | 28 | 31
Percentage of participants
  Omicron (BA.4/BA.5)- Neutralizing Titers | 67.9 [47.6 to 84.1] | 85.2 [66.3 to 95.8] | 42.9 [24.5 to 62.8] | 74.2 [55.4 to 88.1]
  Reference-Strain Neutralizing Titers | 46.4 [27.5 to 66.1] | 63.0 [42.4 to 80.6] | 32.1 [15.9 to 52.4] | 48.4 [30.2 to 66.9]

42. Secondary Outcome: SSA: Percentage of Participants With Seroresponse Based on SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers at 4 Weeks After Vaccination (>=65 Years)
Description: as for outcome 41
Time Frame: SSA:4 Weeks after Vaccination
Population: as for outcome 37
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV
Number analyzed (Participants) | 32 | 32 | 32 | 32
Percentage of participants
  Omicron (BA.4/BA.5)- Neutralizing Titers | 34.4 [18.6 to 53.2] | 28.1 [13.7 to 46.7] | 35.5 [19.2 to 54.6] | 25.0 [11.5 to 43.4]
  Reference-Strain Neutralizing Titers | 21.9 [9.3 to 40.0] | 15.6 [5.3 to 32.8] | 25.0 [11.5 to 43.4] | 18.8 [7.2 to 36.4]

43. Secondary Outcome: SSB: GMTs of Strain-Specific HAI Before Vaccination and at 4 Weeks After Vaccination (18- 64 Years)
Description: GMTs and 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the concentrations and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria, A/Cambodia and B/Phuket.
Time Frame: SSB: Before Vaccination and 4 Weeks after Vaccination
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 28 | 32 | 122 | 118 | 109 | 28 | 26 | 32 | 29 | 26 | 30 | 25
Titers
  A/Wisconsin: Before vaccination: number analyzed (Participants) | 28 | 32 | 120 | 118 | 107 | 28 | 26 | 32 | 28 | 26 | 29 | 25
  A/Wisconsin: Before vaccination | 51.2 [27.2 to 96.6] | 44.6 [26.4 to 75.3] | 44.4 [35.0 to 56.2] | 53.3 [41.1 to 69.2] | 53.5 [41.9 to 68.4] | 46.4 [30.4 to 70.8] | 55.1 [33.3 to 91.0] | 51.9 [33.2 to 81.2] | 45.3 [29.9 to 68.5] | 31.5 [17.8 to 55.7] | 46.2 [26.6 to 80.2] | 37.8 [21.2 to 67.4]
  A/Wisconsin: 4 Weeks after vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 108 | 28 | 26 | 32 | 29 | 25 | 29 | 25
  A/Wisconsin: 4 Weeks after vaccination | 181.1 [114.0 to 287.7] | 343.9 [232.1 to 509.5] | 213.4 [171.8 to 265.1] | 277.3 [228.1 to 337.1] | 215.8 [175.0 to 266.3] | 217.1 [137.2 to 343.4] | 155.8 [98.5 to 246.3] | 149.9 [103.3 to 217.5] | 120.1 [87.3 to 165.3] | 139.3 [90.7 to 213.9] | 173.2 [112.6 to 266.4] | 178.8 [114.0 to 280.4]
  A/Darwin: Before vaccination: number analyzed (Participants) | 27 | 32 | 121 | 118 | 108 | 27 | 26 | 32 | 28 | 25 | 28 | 25
  A/Darwin: Before vaccination | 33.7 [18.5 to 61.4] | 35.1 [23.0 to 53.6] | 22.6 [18.8 to 27.1] | 36.2 [29.3 to 44.7] | 31.3 [25.9 to 38.0] | 51.7 [32.5 to 82.2] | 62.9 [41.7 to 94.9] | 31.5 [22.1 to 45.0] | 38.1 [26.4 to 54.8] | 18.4 [11.3 to 30.1] | 26.9 [16.2 to 44.8] | 18.9 [11.9 to 30.2]
  A/Darwin: 4 Weeks after vaccination: number analyzed (Participants) | 27 | 31 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 25 | 28 | 25
  A/Darwin: 4 Weeks after vaccination | 82.1 [51.9 to 129.9] | 172.3 [126.4 to 235.0] | 110.0 [90.4 to 134.0] | 173.4 [142.9 to 210.3] | 149.6 [121.6 to 184.1] | 172.3 [112.3 to 264.6] | 125.9 [88.4 to 179.3] | 110.7 [83.4 to 147.0] | 106.6 [80.0 to 141.9] | 80.0 [52.9 to 120.9] | 141.4 [96.0 to 208.3] | 99.9 [68.6 to 145.4]
  B/Austria: Before vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 108 | 28 | 26 | 32 | 29 | 26 | 29 | 25
  B/Austria: Before vaccination | 21.0 [11.6 to 38.1] | 13.3 [8.5 to 20.6] | 17.3 [13.9 to 21.6] | 19.2 [15.3 to 24.1] | 20.1 [15.9 to 25.4] | 14.9 [9.7 to 22.7] | 33.2 [19.7 to 56.0] | 12.2 [8.4 to 17.6] | 20.0 [13.1 to 30.5] | 12.7 [8.4 to 19.3] | 16.9 [10.8 to 26.5] | 16.0 [9.4 to 27.3]
  B/Austria: 4 Weeks after vaccination: number analyzed (Participants) | 28 | 31 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 26 | 29 | 25
  B/Austria: 4 Weeks after vaccination | 36.2 [22.7 to 57.8] | 37.4 [24.7 to 56.8] | 32.2 [25.9 to 40.0] | 33.1 [26.6 to 41.3] | 30.7 [24.6 to 38.3] | 26.9 [16.9 to 42.9] | 66.4 [43.5 to 101.4] | 22.3 [15.1 to 32.8] | 28.6 [19.5 to 42.0] | 23.5 [15.4 to 35.8] | 36.4 [23.1 to 57.3] | 27.1 [16.5 to 44.6]
  B/Phuket: Before vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 106 | 28 | 26 | 32 | 29 | 0 | 0 | 25
  B/Phuket: Before vaccination | 35.3 [24.3 to 51.3] | 26.5 [17.2 to 40.9] | 24.0 [19.7 to 29.3] | 25.3 [20.9 to 30.6] | 25.6 [21.1 to 31.2] | 18.6 [12.4 to 27.8] | 20.0 [13.1 to 30.6] | 23.3 [15.3 to 35.4] | 15.0 [10.4 to 21.6] |  |  | 18.4 [12.1 to 27.9]
  B/Phuket: 4 Weeks after vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 106 | 28 | 26 | 32 | 29 | 0 | 0 | 24
  B/Phuket: 4 Weeks after vaccination | 52.5 [36.6 to 75.3] | 49.7 [32.1 to 76.9] | 44.3 [36.0 to 54.7] | 48.0 [40.0 to 57.6] | 46.2 [38.6 to 55.3] | 27.6 [18.8 to 40.5] | 36.0 [22.1 to 58.5] | 46.5 [32.6 to 66.6] | 23.1 [15.6 to 34.3] |  |  | 38.9 [24.7 to 61.1]
  A/Cambodia: Before vaccination: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 18
  A/Cambodia: Before vaccination |  |  |  |  |  |  |  |  |  | 13.1 [8.3 to 20.4] |  | 27.2 [15.8 to 46.9]
  A/Cambodia: 4 Weeks after vaccination: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 0 | 24
  A/Cambodia: 4 Weeks after vaccination |  |  |  |  |  |  |  |  |  | 60.6 [40.5 to 90.9] |  | 77.7 [60.5 to 99.9]

44. Secondary Outcome: SSB: GMFR of Strain-Specific HAI From Before Vaccination to 4 Weeks After Vaccination (18- 64 Years)
Description: GMFRs and the corresponding 2-sided 95% CIs were calculated by exponentiating the mean logarithm of the fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the LLOQ were set to 0.5*LLOQ. When pre-vaccination assay results were lower than the LLOQ and the post-vaccination results were greater than or equal to the LLOQ, the pre-vaccination assay results were set to LLOQ for the GMFR calculation. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria, A/Cambodia and B/Phuket.
Time Frame: SSB: Before Vaccination to 4 Weeks after Vaccination
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: Fold Rise
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 28 | 32 | 122 | 118 | 109 | 28 | 26 | 32 | 29 | 26 | 30 | 25
Fold Rise
  A/Wisconsin: number analyzed (Participants) | 28 | 32 | 120 | 118 | 107 | 28 | 26 | 32 | 28 | 25 | 29 | 25
  A/Wisconsin | 3.1 [1.9 to 5.3] | 6.9 [4.1 to 11.7] | 4.5 [3.7 to 5.5] | 4.8 [3.8 to 5.9] | 3.8 [3.1 to 4.7] | 4.5 [2.8 to 7.1] | 2.8 [1.8 to 4.3] | 2.7 [2.1 to 3.4] | 2.4 [1.7 to 3.6] | 3.6 [2.3 to 5.5] | 3.5 [2.4 to 5.1] | 4.0 [3.0 to 5.4]
  A/Darwin: number analyzed (Participants) | 27 | 31 | 121 | 118 | 107 | 27 | 26 | 32 | 28 | 24 | 27 | 25
  A/Darwin | 2.3 [1.4 to 3.7] | 4.2 [2.9 to 6.1] | 4.4 [3.7 to 5.2] | 4.4 [3.6 to 5.3] | 4.4 [3.6 to 5.4] | 3.5 [2.3 to 5.4] | 1.9 [1.4 to 2.8] | 3.3 [2.5 to 4.4] | 2.8 [2.0 to 4.1] | 3.3 [2.4 to 4.4] | 4.7 [3.3 to 6.5] | 4.3 [3.1 to 6.0]
  B/Austria: number analyzed (Participants) | 28 | 31 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 26 | 29 | 25
  B/Austria | 1.3 [1.0 to 1.8] | 2.2 [1.6 to 3.0] | 1.6 [1.4 to 1.8] | 1.5 [1.4 to 1.7] | 1.4 [1.3 to 1.6] | 1.6 [1.3 to 2.0] | 1.8 [1.4 to 2.5] | 1.6 [1.3 to 2.0] | 1.3 [1.0 to 1.6] | 1.6 [1.3 to 2.0] | 1.9 [1.4 to 2.6] | 1.4 [1.2 to 1.6]
  B/Phuket: number analyzed (Participants) | 28 | 32 | 121 | 118 | 106 | 28 | 26 | 32 | 29 | 0 | 0 | 24
  B/Phuket | 1.4 [1.1 to 1.9] | 1.8 [1.3 to 2.4] | 1.7 [1.5 to 1.9] | 1.8 [1.6 to 2.0] | 1.7 [1.5 to 2.0] | 1.3 [1.1 to 1.6] | 1.7 [1.4 to 2.1] | 1.7 [1.5 to 2.0] | 1.4 [1.1 to 1.7] |  |  | 1.8 [1.5 to 2.3]
  A/Cambodia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 0 | 17
  A/Cambodia |  |  |  |  |  |  |  |  |  | 3.5 [2.5 to 4.9] |  | 2.4 [1.8 to 3.2]

45. Secondary Outcome: SSB: Percentage of Participants Achieving HAI Seroconversion for Each Strain at 4 Weeks After Vaccination (18- 64 Years)
Description: Seroconversion was defined as an HAI titer <1:10 prior to vaccination and >=1:40 at the time point of interest, or an HAI titer of >=1:10 prior to vaccination with a 4-fold rise at the time point of interest. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria,
Time Frame: SSB: 4 Weeks after Vaccination
Population: EIP included all eligible participants who receive study intervention to which they were randomized;had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations."Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. And 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 28 | 32 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 26 | 29 | 25
Percentage of participants
  A/Wisconsin: number analyzed (Participants) | 28 | 32 | 120 | 118 | 107 | 28 | 26 | 32 | 29 | 25 | 29 | 25
  A/Wisconsin | 42.9 [24.5 to 62.8] | 65.6 [46.8 to 81.4] | 64.2 [54.9 to 72.7] | 62.7 [53.3 to 71.4] | 56.1 [46.1 to 65.7] | 64.3 [44.1 to 81.4] | 34.6 [17.2 to 55.7] | 34.4 [18.6 to 53.2] | 25.0 [10.7 to 44.9] | 40.0 [21.1 to 61.3] | 44.8 [26.4 to 64.3] | 68.0 [46.5 to 85.1]
  A/Darwin: number analyzed (Participants) | 27 | 31 | 121 | 118 | 107 | 27 | 26 | 32 | 28 | 24 | 27 | 25
  A/Darwin | 40.7 [22.4 to 61.2] | 61.3 [42.2 to 78.2] | 64.5 [55.2 to 73.0] | 64.4 [55.1 to 73.0] | 64.5 [54.6 to 73.5] | 59.3 [38.8 to 77.6] | 19.2 [6.6 to 39.4] | 56.3 [37.7 to 73.6] | 39.3 [21.5 to 59.4] | 50.0 [29.1 to 70.9] | 70.4 [49.8 to 86.2] | 64.0 [42.5 to 82.0]
  A/Cambodia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 25 | 0 | 17
  A/Cambodia |  |  |  |  |  |  |  |  |  | 60.0 [38.7 to 78.9] |  | 35.3 [14.2 to 61.7]
  B/Austria: number analyzed (Participants) | 28 | 31 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 26 | 29 | 25
  B/Austria | 17.9 [6.1 to 36.9] | 25.8 [11.9 to 44.6] | 16.5 [10.4 to 24.4] | 12.7 [7.3 to 20.1] | 9.3 [4.6 to 16.5] | 14.3 [4.0 to 32.7] | 23.1 [9.0 to 43.6] | 21.9 [9.3 to 40.0] | 10.3 [2.2 to 27.4] | 15.4 [4.4 to 34.9] | 20.7 [8.0 to 39.7] | 4.0 [0.1 to 20.4]
  B/Phuket: number analyzed (Participants) | 28 | 32 | 121 | 118 | 106 | 28 | 26 | 32 | 29 | 0 | 0 | 24
  B/Phuket | 7.1 [0.9 to 23.5] | 25.0 [11.5 to 43.4] | 14.9 [9.1 to 22.5] | 18.6 [12.1 to 26.9] | 14.2 [8.1 to 22.3] | 7.1 [0.9 to 23.5] | 11.5 [2.4 to 30.2] | 6.3 [0.8 to 20.8] | 13.8 [3.9 to 31.7] |  |  | 16.7 [4.7 to 37.4]

46. Secondary Outcome: SSB: Percentage of Participants With Strain Specific HAI Titers >=1:40 Before Vaccination and at 4 Weeks After Vaccination (18- 64 Years)
Description: Percentage of participants with HAI titer >=1:40 for each strain before vaccination and 4 weeks after vaccination is presented in this outcome measure. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Data is reported for following strains: A/Wisconsin, A/Darwin, B/Austria, A/Cambodia and B/Phuket.
Time Frame: SSB: Before Vaccination and at 4 Weeks after Vaccination
Population: EIP included all eligible participants who received vaccination 1; had blood drawn for assay testing within the specified time frame after vaccination; had at least 1 valid and determinate assay result at the 4-week post-vaccination visit and had no major protocol deviations before vaccination. "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here, 'Number Analyzed' signifies number of participants evaluable for the specified rows.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
Number analyzed (Participants) | 28 | 32 | 121 | 118 | 108 | 28 | 26 | 32 | 29 | 26 | 29 | 25
Percentage of participants
  A/Wisconsin: Before Vaccination: number analyzed (Participants) | 28 | 32 | 120 | 118 | 107 | 28 | 26 | 32 | 28 | 26 | 29 | 25
  A/Wisconsin: Before Vaccination | 64.3 [44.1 to 81.4] | 65.6 [46.8 to 81.4] | 64.2 [54.9 to 72.7] | 69.5 [60.3 to 77.6] | 71.0 [61.5 to 79.4] | 71.4 [51.3 to 86.8] | 61.5 [40.6 to 79.8] | 78.1 [60.0 to 90.7] | 71.4 [51.3 to 86.8] | 50.0 [29.9 to 70.1] | 65.5 [45.7 to 82.1] | 64.0 [42.5 to 82.0]
  A/Wisconsin: 4 weeks after vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 108 | 28 | 26 | 32 | 29 | 25 | 29 | 25
  A/Wisconsin: 4 weeks after vaccination | 92.9 [76.5 to 99.1] | 100.0 [89.1 to 100.0] | 95.0 [89.5 to 98.2] | 99.2 [95.4 to 100.0] | 97.2 [92.1 to 99.4] | 96.4 [81.7 to 99.9] | 96.2 [80.4 to 99.9] | 93.8 [79.2 to 99.2] | 96.6 [82.2 to 99.9] | 88.0 [68.8 to 97.5] | 89.7 [72.6 to 97.8] | 92.0 [74.0 to 99.0]
  A/Darwin: Before Vaccination: number analyzed (Participants) | 27 | 32 | 121 | 118 | 108 | 27 | 26 | 32 | 28 | 25 | 28 | 25
  A/Darwin: Before Vaccination | 40.7 [22.4 to 61.2] | 62.5 [43.7 to 78.9] | 45.5 [36.4 to 54.8] | 64.4 [55.1 to 73.0] | 61.1 [51.3 to 70.3] | 74.1 [53.7 to 88.9] | 84.6 [65.1 to 95.6] | 56.3 [37.7 to 73.6] | 67.9 [47.6 to 84.1] | 44.0 [24.4 to 65.1] | 46.4 [27.5 to 66.1] | 44.0 [24.4 to 65.1]
  A/Darwin: 4 weeks after vaccination: number analyzed (Participants) | 27 | 31 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 25 | 28 | 25
  A/Darwin: 4 weeks after vaccination | 81.5 [61.9 to 93.7] | 100.0 [88.8 to 100.0] | 92.6 [86.3 to 96.5] | 96.6 [91.5 to 99.1] | 95.3 [89.4 to 98.5] | 92.9 [76.5 to 99.1] | 96.2 [80.4 to 99.9] | 96.9 [83.8 to 99.9] | 96.6 [82.2 to 99.9] | 88.0 [68.8 to 97.5] | 92.9 [76.5 to 99.1] | 88.0 [68.8 to 97.5]
  A/Cambodia: Before Vaccination: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 26 | 0 | 25
  A/Cambodia: Before Vaccination |  |  |  |  |  |  |  |  |  | 30.8 [14.3 to 51.8] |  | 61.1 [35.7 to 82.7]
  A/Cambodia: 4 weeks after vaccination: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 0 | 24
  A/Cambodia: 4 weeks after vaccination |  |  |  |  |  |  |  |  |  | 88.0 [68.8 to 97.5] |  | 91.7 [73.0 to 99.0]
  B/Austria: Before Vaccination | 42.9 [24.5 to 62.8] | 25.0 [11.5 to 43.4] | 30.6 [22.5 to 39.6] | 33.9 [25.4 to 43.2] | 32.4 [23.7 to 42.1] | 39.3 [21.5 to 59.4] | 50.0 [29.9 to 70.1] | 15.6 [5.3 to 32.8] | 41.4 [23.5 to 61.1] | 19.2 [6.6 to 39.4] | 31.0 [15.3 to 50.8] | 36.0 [18.0 to 57.5]
  B/Austria: 4 weeks after vaccination: number analyzed (Participants) | 28 | 31 | 121 | 118 | 107 | 28 | 26 | 32 | 29 | 26 | 29 | 25
  B/Austria: 4 weeks after vaccination | 53.6 [33.9 to 72.5] | 58.1 [39.1 to 75.5] | 55.4 [46.1 to 64.4] | 53.4 [44.0 to 62.6] | 52.3 [42.5 to 62.1] | 53.6 [33.9 to 72.5] | 80.8 [60.6 to 93.4] | 40.6 [23.7 to 59.4] | 55.2 [35.7 to 73.6] | 34.6 [17.2 to 55.7] | 58.6 [38.9 to 76.5] | 48.0 [27.8 to 68.7]
  B/Phuket: Before Vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 106 | 28 | 26 | 32 | 29 | 0 | 0 | 25
  B/Phuket: Before Vaccination | 60.7 [40.6 to 78.5] | 43.8 [26.4 to 62.3] | 44.6 [35.6 to 53.9] | 45.8 [36.6 to 55.2] | 43.4 [33.8 to 53.4] | 39.3 [21.5 to 59.4] | 34.6 [17.2 to 55.7] | 50.0 [31.9 to 68.1] | 31.0 [15.3 to 50.8] |  |  | 44.0 [24.4 to 65.1]
  B/Phuket: 4 weeks after vaccination: number analyzed (Participants) | 28 | 32 | 121 | 118 | 106 | 28 | 26 | 32 | 29 | 0 | 0 | 24
  B/Phuket: 4 weeks after vaccination | 78.6 [59.0 to 91.7] | 68.8 [50.0 to 83.9] | 61.2 [51.9 to 69.9] | 72.0 [63.0 to 79.9] | 70.8 [61.1 to 79.2] | 50.0 [30.6 to 69.4] | 53.8 [33.4 to 73.4] | 68.8 [50.0 to 83.9] | 41.4 [23.5 to 61.1] |  |  | 58.3 [36.6 to 77.9]

47. Secondary Outcome: SSB: GMTs of SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers Before Vaccination and at 4 Weeks After Vaccination (18- 64 Years)
Description: as for outcome 38
Time Frame: SSB: Before Vaccination and at 4 Weeks after Vaccination
Population: EIP included all eligible participants who receive study intervention to which they were randomized;had blood drawn for assay testing within specified time frame after vaccination;had at least 1 valid & determinate assay result at 4-week post-vaccination visit & had no major protocol deviations."Number of Participants Analyzed" =participants evaluable & 'Number Analyzed' = participants evaluable for specified rows. Only arms which received covid vaccine (BNT162b2) were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg)
Number analyzed (Participants) | 28 | 32 | 122 | 118 | 109 | 28 | 26 | 32 | 29 | 26 | 30
Titers
  Omicron (BA.4/BA.5)- Neutralizing Titers: Before Vaccination: number analyzed (Participants) | 28 | 32 | 120 | 118 | 108 | 27 | 26 | 32 | 28 | 26 | 29
  Omicron (BA.4/BA.5)- Neutralizing Titers: Before Vaccination | 989.5 [524.6 to 1866.2] | 1081.4 [622.6 to 1878.2] | 1127.6 [827.8 to 1535.9] | 1289.6 [997.2 to 1667.7] | 1361.4 [1041.5 to 1779.5] | 1805.5 [1021.6 to 3191.0] | 1527.8 [870.8 to 2680.3] | 1343.6 [887.6 to 2033.9] | 1207.8 [694.2 to 2101.3] | 1688.9 [1064.0 to 2680.7] | 1054.2 [576.3 to 1928.4]
  Omicron (BA.4/BA.5)- Neutralizing Titers: 4 Weeks After Vaccination: number analyzed (Participants) | 28 | 32 | 122 | 117 | 109 | 27 | 26 | 31 | 29 | 26 | 30
  Omicron (BA.4/BA.5)- Neutralizing Titers: 4 Weeks After Vaccination | 4353.8 [2783.5 to 6810.1] | 2960.9 [1867.0 to 4695.9] | 3606.3 [2902.8 to 4480.3] | 3555.6 [2901.5 to 4357.2] | 3997.9 [3197.4 to 4998.8] | 4131.7 [2663.8 to 6408.6] | 3878.7 [2431.9 to 6186.4] | 3999.6 [2780.1 to 5753.9] | 6018.8 [4347.5 to 8332.4] | 4659.7 [3181.4 to 6825.0] | 4385.7 [2546.4 to 7553.6]
  Reference-Strain Neutralizing Titers: Before Vaccination: number analyzed (Participants) | 28 | 32 | 120 | 118 | 108 | 28 | 26 | 32 | 29 | 26 | 28
  Reference-Strain Neutralizing Titers: Before Vaccination | 3396.1 [1798.7 to 6412.1] | 3569.4 [2078.0 to 6131.0] | 4128.9 [3186.9 to 5349.3] | 4335.7 [3490.1 to 5386.1] | 4260.5 [3401.1 to 5337.0] | 4846.4 [3179.9 to 7386.1] | 5693.9 [3566.5 to 9090.3] | 4255.8 [2915.9 to 6211.3] | 4840.6 [3256.3 to 7195.8] | 5380.6 [3260.2 to 8880.2] | 3678.1 [2256.0 to 5996.7]
  Reference-Strain Neutralizing Titers: 4 Weeks After Vaccination: number analyzed (Participants) | 27 | 31 | 121 | 117 | 109 | 27 | 26 | 32 | 29 | 26 | 30
  Reference-Strain Neutralizing Titers: 4 Weeks After Vaccination | 8132.5 [5096.4 to 12977.5] | 7499.8 [5006.7 to 11234.3] | 10769.8 [8913.3 to 13013.1] | 10818.7 [9168.3 to 12766.1] | 12081.5 [9913.1 to 14724.1] | 11319.8 [8175.0 to 15674.2] | 9991.0 [5806.7 to 17190.6] | 11632.2 [8796.5 to 15382.0] | 14921.6 [10784.9 to 20645.0] | 10981.2 [8062.1 to 14957.2] | 14605.4 [9717.6 to 21951.8]

48. Secondary Outcome: SSB: GMFR of SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers From Before Vaccination to 4 Weeks After Vaccination (18- 64 Years)
Description: as for outcome 39
Time Frame: SSB: 4 Weeks after Vaccination
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg)
Number analyzed (Participants) | 28 | 32 | 122 | 118 | 109 | 28 | 26 | 32 | 29 | 26 | 30
Fold rise
  Omicron (BA.4/BA.5)- Neutralizing Titers: number analyzed (Participants) | 28 | 32 | 120 | 117 | 108 | 26 | 26 | 31 | 28 | 26 | 29
  Omicron (BA.4/BA.5)- Neutralizing Titers | 4.1 [2.4 to 6.9] | 2.7 [1.6 to 4.5] | 3.0 [2.5 to 3.7] | 2.6 [2.2 to 3.2] | 2.8 [2.3 to 3.5] | 2.6 [1.8 to 3.7] | 2.5 [1.6 to 3.8] | 2.9 [2.2 to 3.8] | 4.6 [3.0 to 7.0] | 2.8 [1.9 to 4.0] | 3.7 [2.6 to 5.3]
  Reference-Strain Neutralizing Titers: number analyzed (Participants) | 27 | 31 | 119 | 117 | 108 | 27 | 26 | 32 | 29 | 26 | 28
  Reference-Strain Neutralizing Titers | 2.4 [1.5 to 3.8] | 2.1 [1.4 to 3.1] | 2.6 [2.2 to 3.1] | 2.5 [2.1 to 3.0] | 2.8 [2.4 to 3.3] | 2.5 [1.9 to 3.3] | 1.8 [1.0 to 3.1] | 2.7 [2.2 to 3.5] | 3.1 [2.1 to 4.5] | 2.0 [1.2 to 3.5] | 3.8 [2.6 to 5.6]

49. Secondary Outcome: SSB: Percentage of Participants With Seroresponse Based on SARS-CoV-2 Omicron (BA.4/BA.5)- Neutralizing Titers and SARS-CoV-2-Reference-Strain Neutralizing Titers at 4 Weeks After Vaccination (18- 64 Years)
Description: as for outcome 41
Time Frame: SSB: 4 Weeks after Vaccination
Population: as for outcome 47
Measure: Geometric Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg)
Number analyzed (Participants) | 28 | 32 | 120 | 117 | 108 | 27 | 26 | 32 | 29 | 26 | 29
Percentage of participants
  Omicron (BA.4/BA.5)- Neutralizing Titers: number analyzed (Participants) | 28 | 32 | 120 | 117 | 108 | 26 | 26 | 31 | 28 | 26 | 29
  Omicron (BA.4/BA.5)- Neutralizing Titers | 50.0 [30.6 to 69.4] | 37.5 [21.1 to 56.3] | 35.8 [27.3 to 45.1] | 29.9 [21.8 to 39.1] | 30.6 [22.1 to 40.2] | 38.5 [20.2 to 59.4] | 30.8 [14.3 to 51.8] | 38.7 [21.8 to 57.8] | 46.4 [27.5 to 66.1] | 26.9 [11.6 to 47.8] | 44.8 [26.4 to 64.3]
  Reference-Strain Neutralizing Titers: number analyzed (Participants) | 27 | 31 | 119 | 117 | 108 | 27 | 26 | 32 | 29 | 26 | 28
  Reference-Strain Neutralizing Titers | 33.3 [16.5 to 54.0] | 25.8 [11.9 to 44.6] | 33.6 [25.2 to 42.8] | 30.8 [22.6 to 40.0] | 31.5 [22.9 to 41.1] | 25.9 [11.1 to 46.3] | 23.1 [9.0 to 43.6] | 25.0 [11.5 to 43.4] | 41.4 [23.5 to 61.1] | 23.1 [9.0 to 43.6] | 42.9 [24.5 to 62.8]

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events (Systematic assessment): from Day 1 to Day 7 after vaccination; Non-systematic assessment: All-cause mortality/ SAEs: from vaccination up to 6 months after vaccination: other AEs: from vaccination up to 4 weeks after last vaccination.
Description: Same event may appear as both non-SAE and SAE but are distinct events. An event may be categorized as serious in 1 participant and non-serious in another, or a participant may have experienced both AE and non-SAE. Safety population included all participants who received the study intervention. Participants were analyzed according to the treatment which they received.
Arm/Group | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, 18-64 Years: qIRV 30 mcg | Substudy A, 18-64 Years: qIRV 60 mcg | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy A, >=65 Years: qIRV 30 mcg | Substudy A, >=65 Years: qIRV 60 mcg | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) | Substudy B, 18-64 Years: qIRV (30 mcg)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/28 | 0/30 | 0/30 | 0/30 | 0/32 | 0/33 | 0/32 | 0/33 | 0/33 | 0/33 | 0/33 | 0/29 | 0/32 | 0/124 | 0/122 | 0/114 | 0/31 | 0/30 | 0/33 | 0/30 | 0/26 | 0/32 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/28 | 0/30 | 0/30 | 0/30 | 1/32 | 0/33 | 0/32 | 0/33 | 2/33 | 0/33 | 0/33 | 0/29 | 0/32 | 0/124 | 0/122 | 0/114 | 1/31 | 0/30 | 0/33 | 0/30 | 0/26 | 0/32 | 0/29
Other Adverse Events (participants affected / at risk) | 26/30 | 27/28 | 24/30 | 22/30 | 24/30 | 27/32 | 31/33 | 22/32 | 29/33 | 25/33 | 27/33 | 20/33 | 19/29 | 23/32 | 107/124 | 104/122 | 95/114 | 26/31 | 27/30 | 29/33 | 23/30 | 20/26 | 24/32 | 20/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) (N=30) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg (N=28) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) (N=30) | Substudy A, 18-64 Years: qIRV 30 mcg (N=30) | Substudy A, 18-64 Years: qIRV 60 mcg (N=30) | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV (N=32) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) (N=33) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) (N=32) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) (N=33) | Substudy A, >=65 Years: qIRV 30 mcg (N=33) | Substudy A, >=65 Years: qIRV 60 mcg (N=33) | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV (N=33) | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) (N=29) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) (N=32) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) (N=124) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) (N=122) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) (N=114) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) (N=31) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) (N=30) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) (N=33) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) (N=30) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) (N=26) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) (N=32) | Substudy B, 18-64 Years: qIRV (30 mcg) (N=29)
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) (N=30) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 60 mcg (N=28) | Substudy A, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) (N=30) | Substudy A, 18-64 Years: qIRV 30 mcg (N=30) | Substudy A, 18-64 Years: qIRV 60 mcg (N=30) | Substudy A, 18-64 Years: Bivalent BNT162b2 (30 mcg) /QIV (N=32) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) (N=33) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (60 mcg) (N=32) | Substudy A, >=65 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) (N=33) | Substudy A, >=65 Years: qIRV 30 mcg (N=33) | Substudy A, >=65 Years: qIRV 60 mcg (N=33) | Substudy A, >=65 Years: Bivalent BNT162b2 (30 mcg) /QIV (N=33) | Substudy B, 18-64 Years: QIV and Bivalent BNT162b2 (30 mcg) (N=29) | Substudy B, 18-64 Years: QIV and bIRV /Bivalent BNT162b2 (45mcg) (N=32) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 1) (N=124) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 2) (N=122) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 1) (N=114) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (75 mcg) (N=31) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 3) (N=30) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 2) (N=33) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (90 mcg Combination 4) (N=30) | Substudy B, 18-64 Years: qIRV /Bivalent BNT162b2 (60 mcg Combination 3) (N=26) | Substudy B, 18-64 Years: tIRV /Bivalent BNT162b2 (75 mcg) (N=32) | Substudy B, 18-64 Years: qIRV (30 mcg) (N=29)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chills (CHILLS) (General disorders) | 16 | 14 | 16 | 7 | 10 | 7 | 12 | 7 | 3 | 2 | 10 | 4 | 3 | 9 | 41 | 47 | 38 | 17 | 10 | 11 | 10 | 8 | 10 | 8
Fatigue (FATIGUE) (General disorders) | 15 | 14 | 18 | 10 | 10 | 15 | 23 | 12 | 19 | 11 | 18 | 11 | 12 | 12 | 75 | 80 | 65 | 21 | 20 | 17 | 21 | 16 | 17 | 11
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (REDNESS) (General disorders) | 4 | 3 | 3 | 1 | 0 | 3 | 6 | 2 | 7 | 2 | 2 | 4 | 0 | 6 | 13 | 22 | 13 | 3 | 4 | 1 | 2 | 4 | 6 | 2
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site pain (PAIN) (General disorders) | 25 | 25 | 24 | 19 | 22 | 23 | 28 | 17 | 27 | 21 | 24 | 16 | 17 | 23 | 95 | 98 | 85 | 25 | 24 | 27 | 20 | 18 | 23 | 20
Injection site swelling (SWELLING) (General disorders) | 5 | 1 | 2 | 1 | 2 | 3 | 3 | 2 | 4 | 2 | 1 | 3 | 1 | 2 | 13 | 18 | 14 | 6 | 4 | 2 | 0 | 3 | 8 | 2
Pyrexia (FEVER) (General disorders) | 4 | 3 | 8 | 4 | 3 | 1 | 2 | 3 | 0 | 1 | 4 | 0 | 1 | 2 | 16 | 22 | 11 | 10 | 3 | 2 | 6 | 2 | 4 | 3
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 4 | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 3 | 0 | 1 | 3 | 2 | 1 | 12 | 8 | 11 | 3 | 3 | 6 | 3 | 3 | 3 | 2
Vomiting (VOMITING) (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 7 | 4 | 0 | 1 | 0 | 0 | 2 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 5 | 5 | 10 | 1 | 4 | 8 | 3 | 1 | 3 | 2 | 5 | 0 | 3 | 3 | 34 | 29 | 28 | 6 | 4 | 7 | 4 | 8 | 5 | 4
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 14 | 9 | 10 | 5 | 5 | 11 | 8 | 4 | 12 | 5 | 8 | 0 | 6 | 8 | 45 | 45 | 38 | 17 | 7 | 11 | 10 | 8 | 13 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (HEADACHE) (Nervous system disorders) | 16 | 16 | 15 | 7 | 12 | 16 | 16 | 6 | 12 | 8 | 7 | 6 | 6 | 12 | 62 | 61 | 48 | 18 | 14 | 13 | 10 | 10 | 15 | 7
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (or its agents) has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT05596734/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-19): https://cdn.clinicaltrials.gov/large-docs/34/NCT05596734/SAP_001.pdf